CLINICAL TRIAL: NCT00325312
Title: Evaluation of the Efficacy of Subcutaneous Carbon Dioxide Insufflations for Treating Acute Non Specific Neck Pain in General Practice
Brief Title: Subcutaneous Carbon Dioxide Insufflations for Acute Non Specific Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forschungsinstitut für Balneologie und Kurortwissenschaft Bad Elster (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-2
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2006-05

CONDITIONS: Neck Pain
Keywords: Neck Pain; Complementary Therapies; Subcutaneous Carbon Dioxide Insufflations; Acute Treatment
MeSH Terms: conditions — Neck Pain | interventions — Carbon Dioxide

INTERVENTIONS:
Drug: carbon dioxide, subcutaneous application

SUMMARY:
The purpose of the trial is to evaluate whether patients with acute non specific neck pain get pain free sooner, if treated with subcutaneous carbon dioxide insufflations compared to sham ultrasound.

DETAILED DESCRIPTION:
Subcutaneous carbon dioxide insufflations popular in Central und Eastern Europe are a safe and inexpensive treatment modality in complementary medicine and are used mainly in musculoskeletal pain and vascular conditions. However, no rigorous trial exists on their efficacy.

The study is designed as a double blind sham controlled randomized trial to evaluate whether patients with acute non specific neck pain get pain free sooner, if treated with subcutaneous carbon dioxide insufflations compared to sham ultrasound.Since acute non specific neck pain is often self limiting, speed of recovery rather than outcome at fixed points in time is evaluated.

Participants receive either a maximum number of 9 subcutaneous carbon dioxide insufflations or a maximum number of 9 sham ultrasound administered by 4 therapists in a randomized order, thrice weekly. Carbon dioxide gas is insufflated subcutaneously at the locations of neck muscle tenderness. Per tender location 25 ml carbon dioxide gas is administered.

Primary outcome measure is recorded daily by means of a diary. Analysis is done by intention to treat. Differences in time curves are tested using the logrank test. Time curves are graphically displayed by a 1 minus survival Kaplan-Meier plot.

ELIGIBILITY:
Inclusion Criteria:

* participants must report neck pain lasting for less than 7 days
* participants must report a current pain intensity of ≥ 40 mm on a 100 mm visual analogue scale.
* participants must state local neck muscles tenderness during clinical examination at one or more locations

Exclusion Criteria:

* neck pain of specific etiology (e.g., radiculopathy, infection, inflammation, primary tumor, or metastases)
* whiplash injury
* former neck surgery
* pregnancy
* breast feeding.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114
Dates: Start 2001-01; Study Completion 2003-03

PRIMARY OUTCOMES:
time to neck pain relief

SECONDARY OUTCOMES:
time to a 50% reduction in pain intensity
affective pain
sensory pain
pain intensity
treatment failure
recurrence of neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brockow, MD, Principal Investigator — FBK Bad Elster
Locations (1):
- Praxis für Allgemeinmedizin Thomas Heißner, Lohmen, Saxony, Germany